CLINICAL TRIAL: NCT02296528
Title: Safety and Efficacy of the Swallow Expansion Device (SED) for Improvement of Swallowing in Patients With Life-threatening Aspiration Secondary to Feeding Tube Dependent Oropharyngeal Dysphagia: A Single-site, Open-label, Phase 1 Human Trial
Brief Title: Safety and Efficacy of the Swallow Expansion Device (SED) for Improvement of Swallowing in Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to close study
Sponsor: Peter Belafsky, MD (Other)
Responsible Party: Sponsor-Investigator, Peter Belafsky, MD, Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 619595
Record Dates: First submitted 2014-11-05; First posted 2014-11-20 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Oropharyngeal Dysphagia (OPD); Dysphagia
Keywords: Feeding Tube Dependent
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Swallowing Expansion Device (Other): Titanium swallowing expansion device
  Interventions: Device: Swallowing Expansion Device

INTERVENTIONS:
Device: Swallowing Expansion Device — SED looks like the letter "T" and has a plate and a post. The plate is like the top part of the "T" or smooth part of the tack. The plate is attached to the cartilage or flexible connective tissue of the throat. The SED post is like the bottom part of the "T" with a small ring. The post permanently sticks out from the throat, like a skin piercing. The SED is made out of titanium because this metal is extremely strong and commonly used in medical devices put into the body, such as hip joints or bone plates.
  Other Names: SED

SUMMARY:
Biomedical devices, such as artificial joints and pacemakers, are accepted and commonly used in medicine. While great progress in biomedical devices has been made for many other disorders, there is currently no device available to assist with the act of deglutition. The investigators have developed a biomedical device (Swallow Expansion Device, SED) that assists with swallowing by mechanically opening the upper esophageal sphincter and allowing food and liquid to safely enter the esophagus. The SED has proven safe in cadaver and live animal studies (Belafsky, 2010).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate if the SED can safely and effectively improve swallowing. Many people with severe swallowing disability (dysphagia) cannot open their upper esophageal sphincter, which is a circular band of muscle that acts like a valve, allowing food to enter the esophagus (food pipe) and go down into the stomach. People with extreme dysphagia may cough and choke on food, liquid, and even their own saliva. These people are always at risk of food/liquid/saliva accidently entering their lungs. This can cause pneumonia and, in some cases, death. The SED was developed by the University of California, Davis, to improve swallowing. The idea for the SED began when 6 people, who had feeding tubes for 100% of their nutrition because of severe swallowing disability, had a long suture thread attached to their throat. Patients pulled the two ends of the suture thread forward and were able to open their upper esophageal sphincter. In fact, their swallowing improved so much that 3 patients went home with the suture in place so that they could eat by mouth. Unfortunately, the skin around the suture became red and painful within 2-9 days of use. The suture was removed, but the idea for the SED was born. Since the suture study, three different models of the SED have been developed, with each subsequent model better able to improve swallowing, patient safety and use with other common medical tests. The current SED model looks like the letter "T" or a office tack used to stick paper on a wall or board. The SED has a plate and a post. The plate is like the top part of the "T" or smooth part of the tack. The plate is attached to the cartilage or flexible connective tissue of the throat. The SED post is like the bottom part of the "T" or pointy part of the tack, but instead of ending with a point, the end has a small ring. The post permanently sticks out from the throat, like a skin piercing, after the neck skin heals over the plate. Healing takes about 8 weeks. The SED is made out of titanium because this metal is extremely strong and commonly used in medical devices put into the body, such as hip joints or bone plates. A person can eat with the SED by having food enter their esophagus when the SED post is pulled forward with their fingers on the ring. Both sheep and human cadaver studies have shown that the SED works extremely well to widely open the upper esophageal sphincter. The University of California, Davis, and the United States Food and Drug Administration (FDA) have determined that the SED is ready to be tested in a small human study.

ELIGIBILITY:
Inclusion Criteria:

* Profound oropharyngeal feeding tube dependent dysphagia of greater than 12 months duration, as documented by the prevalence of aspiration on fluoroscopic swallow study.
* Must be receiving 100% of nutritional requirements by enterogastric tube.
* 18 years of age and older, acceptable forms of documentation for verification of age include birth certificate, passport, and/or driver's license.
* Diminished upper esophageal sphincter opening defined as less than .55 cm for individuals under 65 years of age and less than .40 cm for individuals over 65 years of age on fluoroscopic swallow study.
* Failure of > 3 months of dysphagia therapy within 3 months of study enrollment.
* No documented history of noncompliance with feeding recommendations.
* Cognition that is within normal limits, as evidenced by an Abbreviated Mental Test Score (AMTS) score greater than 6.
* Manual dexterity that is within normal limits for age, sex, and hand, as evaluated by a Block and Box Test (BBT).
* Physical strength to pull the SED forward, as evidenced by the ability to lift a 5 lb weight off of a table and keep it elevated for 10 seconds.
* Ability to understand the informed consent and comply with follow-up, as evidenced by appropriate questions, responses, and comments during the initial evaluations and a normal Abbreviated Mental Test Score.
* Bilateral vocal fold mobility or unilateral vocal fold immobility in which the individual is able to attain complete glottic closure as evidenced on endoscopy.

Exclusion Criteria:

* Profound oropharyngeal feeding tube dependent dysphagia < 12 months duration.
* Esophageal phase dysphagia as defined as personal history and/or documented diagnosis of esophageal dysmotility, hiatal hernia, stricture, eosinophilic esophagitis, erosive peptic esophagitis, and/or systemic disease affecting the esophagus.
* Able to safely consume any food or liquid by mouth, as documented by fluoroscopic swallow study.
* Normal UES opening, as evidenced by UES opening greater than .55 cm for individuals under 65 years of age and greater than .40 cm for individuals over 65 years of age on fluoroscopic swallow study.
* Currently pregnant, as evidenced by a positive result on a pregnancy test if the patient is within child bearing age (younger than 60 years of age).
* 17 years of age and younger, acceptable forms of documentation for verification of age include birth certificate, passport, and/or license.
* Success full receipt of dysphagia therapy or < 3 months of dysphagia therapy within 3 months of study enrollment.
* Lack of manual dexterity to operate swallowing expansion device as determined by a Block and Box Test (BBT) score below the normal limits per age, sex, and hand.
* Inability to lift a 5 lb weight off of a table and keep it elevated for 10 seconds.
* Lack of cognitive ability to operate swallowing expansion device or provide informed consent as evidenced by an Abbreviated Mental Test Score (AMTS) score less than 6.
* Active tumor involving the cricoid or laryngeal cartilage.
* Known allergic reaction to titanium as evidenced by personal history of allergic or adverse reaction to titanium.
* Infection of cartilage, head, and/or neck at time of evaluation and/or implantation as documented by recent imaging study or abnormal physical examination.
* Presence of a tracheotomy tube or airway obstruction necessitating a tracheotomy tube.
* A documented history of noncompliance with recommendations to take nothing by mouth.
* Patients with an insensate larynx. Laryngeal sensation will be assessed with laryngopharyngeal sensory testing. An insensate larynx is defined as a laryngopharyngeal sensory threshold < 6 mmHg air pulse pressure or a complete absence of the laryngeal adductor reflex on palpation of the arytenoid with a flexible laryngoscope.
* Patients with a current, at the time of evaluation, and/or history of Zenker's diverticulum.
* Patients with sialorrhea at the time of evaluation with or without oral commissure incompetence.
* Patients with profound xerostomia at the time of evaluation.
* Patients with orocutaneous or pharyngocutaneous fistulae at the time of evaluation.
* Patients with a current, at the time of evaluation, and/or history of immunosuppression, as defined by the patient having a diagnosed immunodeficiency disorder or on immunosuppressive medication.
* Patients with a current, at the time of evaluation, and/or history of coagulopathy, as defined by the patient having a diagnosed coagulation disorder or on anticoagulation medication (e.g., baby aspirin, over-the-counter non-steroidal anti-inflammatories, herbal agents, and warfarin, etc.) that cannot be temporarily stopped for the procedure.
* Patients taking sedatives, narcotics, muscle-relaxants, anxiolytics, medical marijuana, alcohol, nicotine, medicinal nicotine, or other mind-altering medications that may affect safe patient use of the swallowing device.
* Patients taking antifibrotic medications.
* Patients with bilateral vocal fold immobility in any position, as evidenced on endoscopy.
* Patients with unilateral vocal fold immobility and unable to attain complete glottic closure, as evidenced on endoscopy.
* Patients with current, at the time of evaluation, and/or documented history of subglottic stenosis, as evidenced on endoscopy.
* Patients with current, at the time of evaluation, and/or documented history of airway obstruction, as evidenced on endoscopy.
* Patients with a life expectancy < 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-06; Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Change in Upper Esophageal Sphincter (UES) Opening | Before implantation, 2 months and 2 years post implantation
  UES opening will be measured via fluoroscopy. A digital still image will be captured at the point of maximum UES opening with and without anterior traction of the SED. The software will be calibrated to the known length of the SED that is visible in the fluoroscopic image. The distance between the anterior and posterior pharyngo-esophageal segment at the point of maximum UES opening will be measured. If swallowing is improved and there is no aspiration, the patient will be taught how to coordinate pulling the SED with the correct amount of force at the appropriate time during swallowing.

SECONDARY OUTCOMES:
Change in Penetration Aspiration Scale (PAS) | Before implantation, 2 months and 2 years post implantation
  Swallowing safety will be assessed with the Penetration Aspiration Scale (PAS) via videofluoroscopy. A scale of 1 indicates a safe swallow (material does not enter the airway). A score of 2-3 indicates mild, 4-5 moderate, and >5-8 indicates severe swallowing disability (material enters the airway, it passes below the vocal folds, and no effort is made to expel it). The patient is initially fed a 1 cc bolus of thin barium. If no aspiration is detected, the patient is then administered a 3 cc and then 20 cc bolus, or largest bolus possible, of barium. If any aspiration is detected at any stage of the study, the procedure is terminated immediately. The PAS will be calculated for the largest swallowed bolus size on fluoroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Department of Otolaryngology, Sacramento, California, United States